CLINICAL TRIAL: NCT03028636
Title: LIBERATE - PRO: An Extended Use Registry to Further Develop Understanding of the Long Term Use of the Eclipse™ System for Fecal Incontinence in Women Via Patient Reported Outcomes
Brief Title: LIBERATE - PRO: Eclipse™ System Registry
Acronym: LIBERATEPRO
Status: Completed | Type: Observational
Sponsor: Pelvalon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CA006
Record Dates: First submitted 2016-12-09; First posted 2017-01-23 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Fecal Incontinence; Bowel Dysfunction; Bowel Incontinence; Accidental Bowel Leakage
Keywords: fecal incontinence; bowel control; accidental bowel leakage; medical device; women's health; vaginal insert; pessary; incontinence; bowel continence; pump
MeSH Terms: conditions — Fecal Incontinence; Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective, open label post market registry to collect Patient Reported Outcomes in an online data capture registry, maintained by Pelvalon, of women with fecal incontinence exiting the LIBERATE study (NCT02428595) continuing to use the Eclipse System for bowel control.

DETAILED DESCRIPTION:
All LIBERATE (NCT02428595) study participants who complete the 12 month visit will be invited to participate in the LIBERATE-PRO post market registry in an effort to obtain additional long term quality of life and economic data. Subjects will be sent an email with a link to the survey(s) or mailed printed surveys depending on chosen survey delivery option to be completed at 3, 6, 9, and 12 months.Baseline will be defined as the baseline value in the LIBERATE study, prior to the insertion of the Eclipse System.

The St. Mark's (Vaizey) Incontinence Severity Score will be used to assess the severity of accidental bowel leakage at 3, 6, 9, and 12 months in comparison to how it was prior to joining the LIBERATE study. The score is based on 7 questions and is a measure of severity of fecal incontinence (FI) symptoms, which has been shown to correlate with improvement in frequency of FI episodes and subjects' perceptions of relief. The composite score calculated from these questions reflects the severity of FI and ranges from 0 (complete continence) to 24 (complete incontinence). The change from baseline score will be calculated at each time point. The average change from baseline score, computed as the mean change from baseline across all completed assessments, will be calculated.

The Patient Global Impression of Improvement (PGI-I) is a validated global index used to rate the response of a condition to a therapy on a scale from 1 (Very much better) to 7 (Very much worse). The PGI-I will be used to assess improvement of accidental bowel leakage at 3, 6, 9, and 12 months in comparison to how it was prior to joining the LIBERATE study. The average PGI-I score, computed as the mean score across all completed assessments, will be calculated.

The FIQOL (Fecal Incontinence Quality of Life Questionnaire will be completed at 12 months. The Fecal Incontinence Quality of Life (FIQOL) scale is a 41-item, validated questionnaire completed by the subject. FIQOL has 4 subscales: lifestyle, coping/behavior, depression/self-perception and embarrassment. Each subscale score ranges from 1 to 5, with 1 indicating a lower functional status of quality of life. FIQOL score will be used to assess the changes in quality of life in each of the subscales in comparison to the same scores prior to joining the LIBERATE study.The change from baseline in each of the 4 subscale scores (lifestyle, coping/behavior, depression/self-perception, embarrassment) will be calculated.

The Eclipse Experience feedback (questions related to perceptions of device comfort, satisfaction with usage and features, and impact on daily activities) will be collected at 3, 6, 9, and 12 months.

All outcomes will be summarized descriptively at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed the 12-month visit in the LIBERATE study (NCT02428595)
* Subject has elected to continue to use the Eclipse System outside of the LIBERATE study
* Subject provides electronic informed consent and HIPAA authorization

Exclusion Criteria:

There are no specific exclusions as this is a data collection registry on a commercially approved product

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects exiting the LIBERATE study who are continuing to use the Eclipse System. Since all of the women in the prior LIBERATE study had to be over the age of 19 to participate in it, this means that all subjects in the registry will be over the age of 19 by default. For information about the LIBERATE study including inclusion/exclusion criteria please see NCT02428595.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gena Dunivan, MD, Principal Investigator — Pelvalon Inc.; University of New Mexico
Locations (1):
- Pelvalon, Inc., Sunnyvale, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: LIBERATE Clinical Trials.gov listing — https://clinicaltrials.gov/ct2/show/NCT02428595
- See also: Pelvalon, Eclipse manufacturer and Study Sponsor, website — http://eclipsesystem.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: Consists of patients who elected to continue treatment after the previous LIBERATE study (NCT02428595). All patients had therefore worn the device for at least 12 months prior to entering this study.
  In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
Period: Overall Study
Arm/Group | All Subjects
Started | 17
Completed | 11
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Consists of patients who elected to continue treatment after the previous LIBERATE study (NCT02428595). All patients had therefore worn the device for at least 12 months prior to entering this study.
  In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
  Surveys were completed at 3, 6, 9, and 12 months during the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17
Menopausal Status [Count of Participants; unit: Participants]
  Pre-menopause | 2
  Peri-menopause | 0
  Post-menopause | 15

OUTCOME MEASURES:

1. Primary Outcome: The St. Mark's (Vaizey) Incontinence Severity Score - Average Change From Baseline Score
Description: The score is based on 7 questions and is a measure of severity of fecal incontinence (FI) symptoms, which has been shown to correlate with improvement in frequency of FI episodes and subjects' perceptions of relief. The score reflects the severity of FI and ranges from 0 (complete continence, better outcome) to 24 (complete incontinence, worse outcome). A reduction in the St. Mark's score is a better outcome. The mean change from baseline score (prior to treatment) will be calculated and reported at 3, 6, and 12 months.
Time Frame: 3, 6, 9, and 12 months
Population: The number analyzed for each time point is the number of participants who provided a survey. Some participants provided surveys for some but not all time points.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | All Subjects
Number analyzed (Participants) | 15
Score on a Scale
  Score at 3 months: number analyzed (Participants) | 12
  Score at 3 months | -6.58 (4.96)
  Score at 6 months | -5.47 (5.58)
  Score at 9 months: number analyzed (Participants) | 14
  Score at 9 months | -7.57 (6.37)
  Score at 12 months: number analyzed (Participants) | 11
  Score at 12 months | -4.64 (6.14)

2. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) - Average Change From Baseline Score
Description: The Patient Global Impression of Improvement (PGI-I) is a validated global index used to rate the response of a condition to a therapy on a scale from 1 (Very much better) to 7 (Very much worse). The PGI-I will be used to assess improvement of accidental bowel leakage at 3, 6, 9, and 12 months in comparison to how it was prior to joining the LIBERATE study. The average PGI-I score, computed as the mean score across all completed assessments, will be calculated.
Time Frame: 3, 6, 9, and 12 months
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects at 3 Months: Consists of patients who elected to continue treatment after the previous LIBERATE study (NCT02428595). All patients had therefore worn the device for at least 12 months prior to entering this study.
  In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
  This arm represents patients who completed surveys 3 months into the study.
- All Subjects at 6 Months: Consists of patients who elected to continue treatment after the previous LIBERATE study (NCT02428595). All patients had therefore worn the device for at least 12 months prior to entering this study.
  In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
  This arm represents patients who completed surveys 6 months into the study.
- All Subjects at 9 Months: Consists of patients who elected to continue treatment after the previous LIBERATE study (NCT02428595). All patients had therefore worn the device for at least 12 months prior to entering this study.
  In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
  This arm represents patients who completed surveys 9 months into the study.
- All Subjects at 12 Months: Consists of patients who elected to continue treatment after the previous LIBERATE study (NCT02428595). All patients had therefore worn the device for at least 12 months prior to entering this study.
  In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
  This arm represents patients who completed surveys 12 months into the study.
Arm/Group | All Subjects at 3 Months | All Subjects at 6 Months | All Subjects at 9 Months | All Subjects at 12 Months
Number analyzed (Participants) | 12 | 15 | 15 | 13
Participants
  Very Much Better (1) | 6 | 6 | 7 | 5
  Much Better (2) | 3 | 5 | 5 | 5
  A Little Better (3) | 2 | 3 | 3 | 2
  No Change (4) | 1 | 1 | 0 | 1
  A Little Worse (5) | 0 | 0 | 0 | 0
  Much Worse (6) | 0 | 0 | 0 | 0
  Very Much Worse (7) | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: The FIQOL (Fecal Incontinence Quality of Life) Questionnaire - Average Change From Baseline Score
Description: The Fecal Incontinence Quality of Life (FIQOL) scale is a 41-item, validated questionnaire completed by the subject. FIQOL has 4 subscales: lifestyle, coping/behavior, depression/self-perception and embarrassment. Each subscale score ranges from 1 to 5, with 1 indicating a lower functional status of quality of life. FIQOL score will be used to assess the changes in quality of life in each of the subscales in comparison to the same scores prior to joining the LIBERATE study.The change from baseline in each of the 4 subscale scores (lifestyle, coping/behavior, depression/self-perception, embarrassment) will be calculated. As higher numbers indicate higher function, a positive change is desirable.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 11
Score on a scale
  Change in Lifestyle Subscale score | .74 (.59)
  Change in Coping/Behavior Subscale score | .87 (.82)
  Change in Depression/Self Perception Subscalescore | .94 (.51)
  Change in Embarrassment Subscale score | .76 (1.03)

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the entirety of the study, for 12 months of patient treatment. Data was collected for a total of 24 months across all patients.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT03028636/Prot_SAP_000.pdf